CLINICAL TRIAL: NCT01162954
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Local Tolerability After Administration of Eye Drop DA-6034 in Healthy Volunteers(Phase I)
Brief Title: Phase I Study to Evaluate the Tolerability of Eye Drop DA-6034 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Jeong-Seong Hong/Assistant Manager, Clinical Development Team 1
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DA6034_DES_I
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Dry Eye Syndrome
Keywords: Eye drop, Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — recoflavone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- DA-6034 (Experimental)
  Interventions: Drug: DA-6034
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DA-6034
  Arms: DA-6034
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, 4-period, cross-over clinical trial. The study is designed to evaluate the safety and local tolerability of DA-6034 upon single and repeated-dose topical application to the both eyes in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 year-old healthy subjects

Exclusion Criteria:

* Presence or history of dry eye or other ocular or systemic diseases
* Corrected visual acuity less than 20/40 in either eye at the screening
* Any eye surgery or laser eye surgery within the past six months
* Intraocular pressure greater than 22 mmHg in either eye at the screening
* Break-up time less than 10 sec with OSDI score corresponding to mild to severe dry eye symptoms in either eye at the screening
* Unanesthetized Schirmer scores <10 mm in either eye at the screening

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Ocular symptomatology, ophthalmologic tests | Single dose: up to 5 days, Multiple dose: up to 15 days

SECONDARY OUTCOMES:
Adverse events, vital signs, physical examinations, ECG findings, clinical laboratory tests, ocular symptomatology, ophthalmologic tests, Unanesthetized Schirmer tests | Single dose: up to 10 days, Multiple dose: up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., M.B.A, Principal Investigator — Clinical Research Institute, Seoul National University Hospital
Locations (1):
- Clinical Research Institue, Seoul National University Hospital, Seoul, Chongno-Gu, Yon-Gon Dong 28, South Korea